CLINICAL TRIAL: NCT06448637
Title: DRUG RELEASING BALL vs. PHARMACOACTIVE STENT IN LARGE VESSELS: MORPHOLOGICAL ANALYSIS AND FUNCTION VASOMOTOR (DEBORA STUDY)
Brief Title: DRUG RELEASING BALL vs. PHARMACOACTIVE STENT IN LARGE VESSELS: MORPHOLOGICAL ANALYSIS AND FUNCTION VASOMOTOR (DEBORA STUDY) IN LARGE VESSELS: MORPHOLOGICAL ANALYSIS AND FUNCTION VASOMOTOR (DEBORA STUDY)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC37-DEBORA
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Drug-coated balloon; Vasomotor function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Coated Balloon (DCB) (Active Comparator): Drug Coated Balloon (DCB)
  Interventions: Device: Drug Coated Balloon (DCB)
- Drug Eluting Stent (DES) (Experimental): Drug Eluting Stent (DES)
  Interventions: Device: Drug Eluting Stent (DES)

INTERVENTIONS:
Device: Drug Coated Balloon (DCB) — Drug Coated Balloon (DCB) in patients with indication of Percutaneous Coronary Intervention (PCI)
  Arms: Drug Coated Balloon (DCB)
Device: Drug Eluting Stent (DES) — Drug Eluting Stent (DES) in patients with indication of Percutaneous Coronary Intervention (PCI)
  Arms: Drug Eluting Stent (DES)

SUMMARY:
Randomized, controlled, open and multicenter study that analyzes the vasomotor function 8 months after use of the drug-eluting balloon (DCB) vs. drug-eluting stent (DES) in vessels ≥ 3.5 mm

DETAILED DESCRIPTION:
Randomized, controlled, open and multicenter study that analyzes the vasomotor function 8 months after use of the drug-eluting balloon (DCB) vs. drug-eluting stent (DES) in vessels ≥ 3.5 mm

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following conditions are included.

* Patients aged ≥ 18 years and;
* Patients with chronic coronary syndrome, acute coronary syndrome without ST segment elevation or acute coronary syndrome with elevation ST segment in non-culprit lesions 48 hours after the event and;
* Patients with de novo lesions in vessels ≥ 3.5 mm without calcification significant no visible thrombus and;
* Patients who have been informed of the characteristics of the study and have provided their written informed consent.

Exclusion Criteria:

Patients who meet at least one of the following conditions are excluded:

* Patients with any contraindication for the administration of acetylcholine (ACh) or nitroglycerin (NTG).
* Patients with a history of coronary vasospasm or spontaneous dissection of the coronary artery.
* Patients with significant medical, surgical or psychiatric condition that would affect the safety of the subject or influence the outcome of the study according to the doctor's opinion.
* Patients who received a combination of DES and DCB in the same vessel
* Patients with glomerular filtration rate <30 ml/min/ 1.73 m2
* Patients with body mass index >35 (may affect the evaluation qualitative diameter of the coronary artery).
* Patients with symptomatic congestive heart failure.
* Patients with significant autoimmune inflammatory conditions and patients taking immunomodulatory medications (including methotrexate, cyclosporine, steroids).
* Patients with heart transplant.
* Patients with anemia (Hb <12 g/dL in men and <10 g/dL in women).
* Patients, women of childbearing age with a positive pregnancy test.
* Pregnant female patients.
* Patients included in other clinical trials with active follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of vessels with a positive response to Ach, defined as >4% change in the mean luminal diameter observed in the coronary segment distal (10-30 mm) to the treated segment, after the infusion of the maximum dose of ACh (10-6 mol/L). | 8 months
  Percentage of vessels with a positive response to Ach, defined as >4% change in the mean luminal diameter observed in the coronary segment distal (10-30 mm) to the treated segment, after the infusion of the maximum dose of ACh (10-6 mol/L).

SECONDARY OUTCOMES:
Comparison of percentage of angiographic restenosis by quantitative coronary | 8 months
  Comparison of percentage of angiographic restenosis by quantitative coronary
Comparison of the minimum luminal diameter of the treated segment by optical coronary tomography | 8 months
  Comparison of the minimum luminal diameter of the treated segment by optical coronary tomography
Comparison of the minimum luminal area of the treated segment by optical coronary tomography | 8 months
  Comparison of the minimum luminal area of the treated segment by optical coronary tomography
Percentage of of strut coverage by OCT(Optical Coherence Tomography) in the DES group | 8 months
  Percentage of of strut coverage by OCT in the DES group
Percentage of vessels with normal vascular architecture with correct definition of intima and media by optical coherence tomography in the drug-coated balloon group at 8 months | 8 months
  Percentage of vessels with normal vascular architecture with correct definition of intima and media by optical coherence tomography in the drug-coated balloon group at 8 months

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario de Leon, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Provincial de Pontevedra, Pontevedra

REFERENCES:
- [Background] Yerasi C, Case BC, Forrestal BJ, Torguson R, Weintraub WS, Garcia-Garcia HM, Waksman R. Drug-Coated Balloon for De Novo Coronary Artery Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Mar 10;75(9):1061-1073. doi: 10.1016/j.jacc.2019.12.046. PMID 32138967
- [Background] Nakamura T, Brott BC, Brants I, Panchal D, Li J, Chen JP, King SB 3rd, Chronos N, Hou D. Vasomotor function after paclitaxel-coated balloon post-dilation in porcine coronary stent model. JACC Cardiovasc Interv. 2011 Feb;4(2):247-55. doi: 10.1016/j.jcin.2010.08.028. PMID 21349465
- [Background] Gutierrez E G-LJ, Escaned J, Cruz I, Ojeda S, Romaguera R, Moreno R. Valoración de la función endotelial y provocación de vasoespasmo coronario mediante infusión intracoronaria de acetilcolina. Documento técnico de la ACI-SEC. REC Interv Cardiol. 2021;3(4):286-296.
- [Background] Gomez-Lara J, Oyarzabal L, Ortega-Paz L, Brugaletta S, Romaguera R, Salvatella N, Roura G, Rivero F, Fuentes L, Alfonso F, Otaegui I, Vandeloo B, Vaquerizo B, Sabate M, Comin-Colet J, Gomez-Hospital JA. Coronary Endothelium-Dependent Vasomotor Function After Drug-Eluting Stent and Bioresorbable Scaffold Implantation. J Am Heart Assoc. 2021 Nov 16;10(22):e022123. doi: 10.1161/JAHA.121.022123. Epub 2021 Nov 3. PMID 34729992
- [Background] Brugaletta S, Heo JH, Garcia-Garcia HM, Farooq V, van Geuns RJ, de Bruyne B, Dudek D, Smits PC, Koolen J, McClean D, Dorange C, Veldhof S, Rapoza R, Onuma Y, Bruining N, Ormiston JA, Serruys PW. Endothelial-dependent vasomotion in a coronary segment treated by ABSORB everolimus-eluting bioresorbable vascular scaffold system is related to plaque composition at the time of bioresorption of the polymer: indirect finding of vascular reparative therapy? Eur Heart J. 2012 Jun;33(11):1325-33. doi: 10.1093/eurheartj/ehr466. Epub 2012 Apr 16. PMID 22507972